CLINICAL TRIAL: NCT06491537
Title: Use of Early Time-restricted Eating to Promote Weight Loss and Improve Cardiometabolic Health in Postpartum Women
Brief Title: Time-restricted Eating for Postpartum Weight Loss
Acronym: Time4Mom
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Camille S Worthington, PhD, Primary Investigator, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB-300012535; K23HD108345 (NIH)
Record Dates: First submitted 2024-07-01; First posted 2024-07-09 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Postpartum Weight Retention; Overweight and Obesity
Keywords: postpartum; weight management; time-restricted eating
MeSH Terms: conditions — Gestational Weight Gain; Overweight; Obesity; Intermittent Fasting

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- eTRE Intervention (Experimental): A 9-hour eating/15-hour fasting time-restricted eating (eTRE) intervention with tapered remote behavioral support sessions delivered by a trained interventionist.
  Interventions: Behavioral: Early Time-Restricted Eating (eTRE)
- Control (Active Comparator): Control condition in which participants are instructed to maintain their baseline eating window with tapered remote behavioral support check-ins delivered by a trained interventionist to encourage maintenance of the baseline eating window.
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Early Time-Restricted Eating (eTRE) — 12 weeks of eTRE intervention. Study staff will provide 7 support sessions with brief behavioral support, including evidence based strategies of problem-solving, action planning, and motivational interviewing.
  Other Names: Intermittent Fasting; Timed Eating
  Arms: eTRE Intervention
Behavioral: Control — The control group will be instructed to maintain their average eating window for the 12-week period. Study staff will contact participants 7 times to encourage maintenance.
  Arms: Control

SUMMARY:
This study is being done to assess the feasibility and acceptability of a time-restricted eating intervention among postpartum women with overweight/obesity.

DETAILED DESCRIPTION:
Existing postpartum weight retention (PPWR) interventions have had limited success. Timing-based interventions, such as early time-restricted eating (eTRE), show significant improvements in cardiometabolic endpoints in non-postpartum cohorts. The purpose of the Time4Mom study is to conduct a pilot randomized trial of a postpartum-adapted eTRE intervention to test feasibility and acceptability of the eTRE intervention and trial protocol. We will also compare changes in clinical outcomes of interest and patient-reported outcomes between eTRE (intervention) and control groups.

This 2-arm trial will randomize 60 postpartum women to either Control or eTRE for 12 weeks (n=30/group).

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Experienced a healthy singleton pregnancy
* 6-16 weeks postpartum at enrollment
* Body mass index ≥25 at enrollment
* Willing to consent

Exclusion Criteria:

* Self-reported major health condition (such as renal disease, cancer, or Type 1 or Type 2 diabetes)
* Current treatment for severe psychiatric disorder (such as schizophrenia)
* Self-reported diagnosis of anorexia or bulimia
* Current use of medication expected to significantly impact body weight
* Current substance abuse
* Participation in another dietary and/or weight management intervention postpartum
* Performing overnight shiftwork >1x/week
* Regularly fasting ≥14 hr/day or completing twelve or more 24-hr fasts within the past year
* Unable to understand and communicate in English

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-05-22 (Actual); Primary Completion 2029-01-01 (Estimated); Study Completion 2029-02-01 (Estimated)

PRIMARY OUTCOMES:
Study Participation Rate | Baseline (6-16 weeks postpartum)
  Percentage of eligible subjects who agreed to participate out of those who were screened.
Oral Glucose Tolerance Test (OGTT) | Baseline (6-16 weeks postpartum), follow-up (18-28 weeks postpartum)
  Indices of glucose tolerance and insulin action will be assessed via a 2-hr OGTT. Participants will consume a 75-g glucose load within 5 minutes, which will be timed to begin at each participant's habitual breakfast time. Fasting blood samples will be collected at 15-, 30-, 60-, 90-, and 120-minutes relative to glucose consumption.
Energy Intake | Baseline (6-16 weeks postpartum), follow-up (18-28 weeks postpartum)
  Dietary intake will be collected at each assessment by 3 self-administered 24-hr recalls on 3 non-consecutive days (2 weekdays, 1 weekend day) using the Automatic Self-Administered 24-hour Dietary Assessment Tool (ASA24), an online platform developed and hosted by the National Cancer Institute. Total energy intake and kcals from each macronutrient will be derived from 24-hr recalls.
Participant Retention | Baseline (6-16 weeks postpartum), follow-up (18-28 weeks postpartum)
  The proportion of enrolled participants who complete follow-up.
Change in Visceral Fat | Baseline (6-16 weeks postpartum), follow-up (18-28 weeks postpartum)
  Bioelectrical impedance analysis (BIA) (seca® mBCA 514) will be used to assess visceral adipose tissue.
Participant Adherence to Intervention | Collected daily from intervention start (6-16 weeks postpartum) to follow-up (18-28 weeks postpartum)
  Adherence to eating window based on responses to daily electronic REDCap surveys that record start and stop time of the eating window.
eTRE Intervention Satisfaction | Baseline (6-16 weeks postpartum), follow-up (18-28 weeks postpartum)
  Participant satisfaction with the eating schedule will be assessed using a 5-point Likert scale. Long-term eating schedule preferences will be assessed by asking intervention participants at follow-up whether they plan to: (a) continue following the assigned eTRE schedule; (b) follow a modified eTRE schedule [and specifying what modifications they plan to make]; or (c) stop eTRE and return to prior meal timing habits.
  Qualitative data on eTRE intervention satisfaction will be collected at follow-up. These one-on-one interviews will be conducted in-person or remotely via videoconferencing. Topics explored will include participants' typical day during the intervention, experiences with eTRE, adherence barriers/facilitators, intervention satisfaction, and suggested improvements.
Change in Body Weight | Baseline (6-16 weeks postpartum), follow-up (18-28 weeks postpartum)
  Body weight measured at baseline and follow-up will be used to calculate weight change.
Change in Subjective Appetite | Baseline (6-16 weeks postpartum), follow-up (18-28 weeks postpartum)
  Subjective ratings of appetite (hunger and satiety) over the past week will be collected at baseline and follow-up using visual analogue scales scored from 0 (less hunger/less satiety) to 100 (more feelings of hunger/more feelings of satiety) based on the response along a 100-mm line.
Self-Reported Fatigue | Baseline (6-16 weeks postpartum), follow-up (18-28 weeks postpartum)
  Fatigue will be assessed using the NIH's validated 8-item Patient-Reported Outcomes Measurement Information System (PROMIS) Fatigue Short Form (SF) 8a to assess fatigue over the past 7 days. The PROMIS Fatigue SF 8a is scored on a T-score metric with a mean of 50 and standard deviation of 10. The T-score metric is referenced to the US general population with respect to race/ethnicity, age, education, and sex (e.g., T-score of 40 would be one SD below the US general population). A higher PROMIS T-score represents more of the concept being measured (higher score indicates more fatigue).

CONTACTS AND LOCATIONS:
Overall Officials: Camille Worthington, PhD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: Yes
The following data produced during the project will be preserved and shared: Aggregate data on recruitment rates and reasons for refusal, retention rates, adherence rates, and treatment satisfaction will be shared publicly. Individual participant data (IPD) for the following measures will be restricted with a data use agreement: anthropometrics (weight, height, waist circumference); body composition; the following serum levels at each timepoint from the oral glucose tolerance test: insulin, glucose, and c-peptide; dietary data; survey responses/total scores; demographics; and pregnancy-related medical history.
  All aggregate datasets that can be shared publicly will be deposited in the Open Science Framework (OSF) generalist repository. De-identified IPD will be shared via controlled access in the Vivli repository.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Data will be made available at the time of associated publication or by the end of the clinical trial.
Access Criteria: To request access to the data, the user must submit a valid scientific question, include a statistical analysis plan, and complete all required fields on the Vivli data request form. Vivli will review the data request for completeness. Anyone who has submitted an approved data request and signed a DUA on Vivli will be given access to the data without cost for a set period